CLINICAL TRIAL: NCT02389504
Title: An Investigation of Return to Play Exertion Protocol in Concussed Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary study team member left organization, study was not completed.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Research Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14070006
Record Dates: First submitted 2015-02-26; First posted 2015-03-17 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Concussion
Keywords: Exertion; Efficacy of Treatment
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Physical Therapy Protocol (Active Comparator): Regular Physical Therapy Protocol. Standard treadmill running, monitoring heart rate
  Interventions: Other: Standard Exertional Physical Therapy
- Exertion Physical Therapy Protocol (Experimental): Exertional Physical Therapy Protocol. Dynamic exertion protocol includes the treadmill running aspect, but also incorporates other exercises that involve lateral movement (e.g., side lunges, lateral speed training exercises) as well as planar changes (e.g., burpees, squat thrusts) . Recovery on these exercises is measured based on time subjects are able to tolerate the exertion without symptom increase. Across all exertion protocols additional measures of subjective physical effort and objective measurement of heart rate are taken.
  Interventions: Other: Dynamic Exertional Physical Therapy

INTERVENTIONS:
Other: Dynamic Exertional Physical Therapy — By contrast, the dynamic exertion protocol includes the treadmill running aspect, but also incorporates other exercises that involve lateral movement (e.g., side lunges, lateral speed training exercises) as well as planar changes (e.g., burpees, squat thrusts) . Recovery on these exercises is measured based on time subjects are able to tolerate the exertion without symptom increase. Across all exertion protocols additional measures of subjective physical effort and objective measurement of heart rate are taken.
  Arms: Exertion Physical Therapy Protocol
Other: Standard Exertional Physical Therapy — Standard treadmill running, monitoring heart rate
  Arms: Standard Physical Therapy Protocol

SUMMARY:
An Investigation of Return to Play Exertion Protocol in Concussed Adolescents

DETAILED DESCRIPTION:
Written informed parental consent and assent will be obtained for all subjects. The PI or Co-I will administer ImPACT (Immediate Post-Concussion Assessment and Cognitive Testing), the PCSS (Post Concussion Symptom Scale), and the VOMS (Vestibular Ocular Motor Screening) to each subject during their first clinical visit. In addition to demographic variables such as age and gender, groups will be matched based on ImPACT and VOMS performance as well as the number, type, and severity of symptoms reported on the PCSS. Subjects will be assigned to receive either the currently accepted standard of care (Heart Rate Exertion group) or the newly developed exertion protocol (Dynamic Exertion Group). Participants will be matched according to PCSS total, VOMS symptom report, and by demographic variables including age and gender. The first participant will be assigned to the dynamic exertion group and the next to the standard of care group, alternating accordingly as covariates allow. The physical therapists will be responsible for administering the assigned exertion protocol to each subject across four time points (one week between each session). Follow-up data regarding recovery time (i.e., clinical return to normal activity) will also be collected. Neurocognitive testing will take place on 3-4 week intervals as is consistent with clinical practice. The current study will include a pre-exertion neurocognitive evaluation and a post-exertion protocol neurocognitive evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years of age
* Referred to exertion physical therapy within 6 weeks of sport related concussion

Exclusion Criteria:

* Family history of mood or anxiety disorder
* Diagnosis or treatment of migraine
* Diagnosed history of learning disability, ADHD (Attention Deficit Hyperactivity Disorder)
* Concussion history of 3 or more
* Other factors that would prevent subject from completing exertion protocol

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-20 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the current standard of care exertion protocol versus a newly developed program that emphasizes dynamic movement and sport-specific activities as measured by patient symtom scales and neurocognitive testing performance | 4 weeks
  To empirically assess the efficacy of the current standard of care as it relates to a gradual increase in physical activity relative to a newly developed program. The current standard of care focuses on heart rate and duration of physical activity where all athletes are progressed in the same fashion based on ability to tolerate symptoms while running on a treadmill; by contrast, the newly developed program emphasizes dynamic movement (incorporating lateral movement and planar changes in addition to treadmill running) that more closely approximate movements made while playing sports where rehabilitation is based on specific symptom deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- UMPC Sports Medicine Concussion Research Program, Pittsburgh, Pennsylvania, United States